CLINICAL TRIAL: NCT06392139
Title: A Quasi-experimental Pragmatic Trial Evaluating a Tailored Healthcare Service for Patients With Borderline Personality Disorder: Borderline Personality Disorder Athens Study (BPDAS)
Brief Title: Specialized Healthcare Service for BPD Patients: Athens Trial
Acronym: BPDAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ioannis A. Malogiannis (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University Mental Health Research Institute, Athens, Greece (Other); Sismanogleion General Hospital, 3rd Respiratory Medicine Department (Other); Attikon Hospital (Other)
Responsible Party: Sponsor-Investigator, Ioannis A. Malogiannis, Mr Ioannis A. Malogiannis, Head of the BPD Specific Sector, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. 404/06-07-2021
Record Dates: First submitted 2024-03-06; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Other Mental Conditions
Keywords: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Therapeutics; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): The Specific Therapy Program for Personality Disorders at the 1st Psychiatric Clinic, Medical School, National and Kapodistrian University of Athens, Eginition Hospital, established in 1999, offers outpatient, inpatient, and day care services with psychoanalytic interventions tailored for Borderline Personality Disorder. Group psychoanalytic psychotherapy sessions are predominant, supported by research. Patients undergo initial 6-8 months of closely monitored outpatient care, including monthly psychodynamically oriented sessions, psychiatric appointments, and psychological assessments, focusing on crisis management and personalized treatment plans. Subsequently, long-term psychodynamic psychotherapy interventions, often combined with psychiatric treatment, provide sustained therapeutic support.
  Interventions: Behavioral: Specific Therapy Program for Personality Disorders
- Treatment As Usual (TAU) Group (Active Comparator): The TAU group receives the common practice treatment in the two Specific Outpatient Clinics for BPD patients:
  1. The Outpatient Clinic for Borderline Personality Disorder Patients of the 2nd Psychiatric Clinic at the Medical School of National and Kapodistrian University of Athens called Attikon General University Hospital and
  2. The Outpatient Clinic for Borderline Personality Disorder Patients of the Psychiatric Clinic of Sismanogleion General Hospital.
  Interventions: Other: Treatment As Usual (TAU) Group

INTERVENTIONS:
Behavioral: Specific Therapy Program for Personality Disorders — The program was founded in 1999; since then, it has provided a wide range of different treatment interventions (outpatient, inpatient and day care). The interventions are psychoanalytically oriented and specifically for patients with Borderline Personality Disorder. Most of them are in the form of group psychoanalytic psychotherapy. The program consists of two steps: 1) an initial reception outpatient clinic where patients are followed after the referral to the Program, for a period of 6-8 months. This first step consists of monthly psychodynamically oriented sessions, monthly psychiatric appointments and application of psychological assessment instruments. The intervention focuses on crisis management and construction of the treatment plan for every patient. 2) The second step consists of long-term psychodynamic psychotherapy interventions, in combination with psychiatric treatment when it is is needed.
  Other Names: BPDAS
  Arms: Experimental: Intervention group
Other: Treatment As Usual (TAU) Group — The TAU group receives the common practice treatment in the two Specific Outpatient Clinics for BPD patients:
  The Outpatient Clinic for Borderline Personality Disorder Patients of the 2nd Psychiatric Clinic at the Medical School of National and Kapodistrian University of Athens called Attikon General University Hospital and The Outpatient Clinic for Borderline Personality Disorder Patients of the Psychiatric Clinic of Sismanogleion General Hospital.
  Treatment As Usual (TAU) The TAU includes the psychiatric management, consultation and pharmacotherapy if needed in the two Specific Outpatient Clinics for BPD patients. TAU provides one thirty minutes session per month. In case of crisis management patients contact their psychiatrist during the working hours, or after that they leave a message on the telephone answering machine and if needed make a visit in the Emergency Department of the Hospital on Duty.
  Arms: Treatment As Usual (TAU) Group

SUMMARY:
A quasi-experimental pragmatic trial was developed to evaluate a specific health-care service for the treatment of biporal personality disorder (BPD) patients.The effectiveness and economic evaluation (cost-effectiveness and cost-utility) of this specific health-care service as it is offered in every-day clinical practice will be assesed. The main hypothesis of the particular study is that the specific health-care service for the treatment of BPD patients has better efficacy and cost-effectiveness than the treatment as usual.

Furthermore, two additional substudies will be performed. The first one is a qualitative study on the experiences of patients and therapists of the specific program as compared to common treatment. The second substudy aims to investigate the effectiveness and the possible psychodynamic functions of the initial outpatient reception clinic of the specific program.

Patients will be followed for 2 years.

DETAILED DESCRIPTION:
There is a lack of studies evaluating the effectiveness of health care services providing treatment for patients with borderline personality disorder). This study is the first to evaluate a psychoanalytically-oriented intervention that is developed specifically for BPD.

A quasi-experimental pragmatic trial for the evaluation of a specific health-care service for BPD patients was developed. The effectiveness and economic evaluation (cost-effectiveness and cost-utility) of a special health service for the treatment of BPD patients as it is offered in the every-day clinical practice will be assessed.

This health-care service is the Specific Therapy Program for BPD patients of the 1st Psychiatric Clinic of the Medical School of the National and Kapodistrian University of Athens. It has provided a wide range of different treatment interventions (outpatient, inpatient and day care).

The main hypothesis of the study is that the specific health-care service for the treatment of BPD patients has better efficacy and cost-effectiveness than the treatment as usual.

Furthermore, two additional substudies will be performed. The first one regards a qualitative study on the experiences of patients and therapists of the specific program and of the TAU. Qualitative data will be collected from interviews and/or focus groups. This study aims to provide information on the aspects of the specific health care service that are more advantageous for the patients. The second substudy aims to investigate the effectiveness and the possible psychodynamic functions of the initial outpatient reception clinic of the specific program and will be based both on empirical qualitative data.

Patients will be followed for 2 years. The outcome measures will be assessed at baseline, before the assignment of the patient and every 6 months until the completion of the 2nd year follow-up (6 months, 1 year, 18 months, 2 years). The assessment of the mediators for the evaluation of the mechanisms of change for the patients of the study will be contacted at baseline and then every year (1 year, 2 years). An additional follow up assessment will be administered 6 months and 1 year after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of BPD (diagnosed with Structural Clinical Interview for DSM-5 Personality Disorders; SCID-5-PD and
* willingness to participate in the study.

Exclusion Criteria:

* lifetime psychotic disorder (except for a brief psychotic disorder as described in the Diagnostic and Statistical Manual of Mental Disorders, version V, DSM-5, BPD criterion 9,
* bipolar disorder type I,
* antisocial personality disorder,
* severe substance dependence resulting in severe cognitive restrictions during therapy, needing clinical detoxification,
* IQ below 80,
* organic brain disease,
* poor Greek language skills.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Severity of BPD and severe parasuicidal behavior as defined by Bateman and Fonagy (2009). | Baseline, 6 months, 1 year, 18 months, 2 years
  It is assessed using the Borderline Personality Disorder Severity Index (BPDSI) and the latter is assessed through the number of 1) suicide attempts, 2) life-threatening self-harm behaviors and 3) psychiatric hospital admissions.
Suicide Harm Inventory | Baseline, 6 months, 1 year, 18 months, 2 years
  It is an interview designed to ensure accurate collection of data about attempted acts of suicide and incidents of self-harm over a six-month period but does not aim to measure their severity.

SECONDARY OUTCOMES:
General psychiatric symptoms present at the time of assessment. | Baseline, 6 months, 1 year, 18 months, 2 years
  These will be assessed using the BSI (Brief Symptom Inventory): it is a self-report inventory of general psychiatric symptoms present at the time of assessment.
Subjective Quality of Life | Baseline, 6 months, 1 year, 18 months, 2 years
  It will be assessed using WHOQOL BREF (World Health Organization Quality of Life questionnaire), which is a valid and reliable instrument for the assessment of the quality of life in the two prior weeks. It assesses various domains.
Distress caused by interpersonal problems | Baseline, 6 months, 1 year, 18 months, 2 years
  It will be assessed using the IIP-64 (Inventory of interpersonal problems): it is a 64-item measure designed to determine sources of interpersonal distress.
Functional Impairments in fields such as work and household | Baseline, 6 months, 1 year, 18 months, 2 years
  It will be assessed using WSAS (Work and Social Adjustment Scale): is a self-report instrument that rates functional impairment in the fields of work, household, social leisure, private leisure, family, and relationships.
WHODAS II | Baseline, 6 months, 2 years
  A generic assessment instrument for health and disability.
Reflective Functioning | Baseline,1 year, 2 years
  It will be assessed using the RFQ-8 (Reflective Functioning Questionnaire): is a brief, screening measure of reflective functioning. It has been developed to assess severe impairments or imbalances in mentalizing as typically observed in patients with borderline personality disorder features.
Defense tendency | Baseline,1 year, 2 years
  It will be assessed using DSQ-40 (Defense Style Questionnaire): is a questionnaire of 40 items, aims to assess behavior indicative of conscious derivatives of defensive styles that correspond to hypothesized patterns of unconscious psychological mechanisms.
Personality Organisation | Baseline,1 year, 2 years
  Measured using IPO-GR (Inventory of Personality Organization): it is a self-report instrument intended to measure a patient's level of personality organization.
Client Satisfaction Questionnaire | 6 months, 1 year, 18 months, 2 years
  CSQ-8 The Client Satisfaction Questionnaire (CSQ) is one of the most used questionnaires for measuring patient-reported satisfaction in mental healthcare settings.
Patients' health-related quality of life | Baseline, 6 months, 1 year, 18 months, 2 years
  A five-item self-report measure (EuroQol-5D-3L) will be used to assess five different dimensions of patients' health-related quality of life: self-care, mobility, usual activity, anxiety/depression, and pain/discomfort

OTHER OUTCOMES:
Cost-Effectiveness | Baseline, 6 months, 1 year, 18 months, 2 years
  Αn interview will be conducted to retrospectively identify costs relevant to the experience of patients with BPD. These include health care costs (visits to general practitioners, hospitals, psychiatrists etc.), patient and family costs (travel costs, informal care, out-of-pocket costs, etc.), and costs in other sectors (productivity losses at work, volunteering work, and/or studying, etc.). The recall period for the interview is 6 months.
ALL 3 MECHANISMS OF CHANGE- RFQ, IPO-GR, DSQ-40 | Baseline, 1 year, 2 years
ETI - Early Trauma Inventory | Baseline, 2 years
  The self-report Early Trauma Inventory (ETI-SR-SF) was developed by Bremner et al in 2007 and has been proven a valid tool for the assessment of childhood trauma. The inventory covers four types of traumatic experiences: general trauma, physical abuse, emotional abuse and sexual abuse.

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - 1st Psychiatric Clinic, Medical School, National Kapodistrian University of Athens, Eginition Hospital, Athens, Attica
  - Outpatient Clinic for Borderline Personality Disorder Patients, 2nd Psychiatric Clinic, Medical School of National Kapodistrian University of Athens: Attikon General University Hospital, Athens, Attica
  - Outpatient Clinic for Borderline Personality Disorder Patients, Psychiatric Clinic of Sismanogleion General Hospital, Athens, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Collaborating Centre for Mental Health (UK). Borderline Personality Disorder: Treatment and Management. Leicester (UK): British Psychological Society (UK); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK55403/ PMID 21796831
- [Background] Vaslamatzis G, Coccossis M, Zervis C, Panagiotopoulou V, Chatziandreou M. A psychoanalytically oriented combined treatment approach for severely disturbed borderline patients: the Athens project. Bull Menninger Clin. 2004 Fall;68(4):337-49. doi: 10.1521/bumc.68.4.337.56640. PMID 15843180
- [Background] Vaslamatzis G, Theodoropoulos P, Vondikaki S, Karamanolaki H, MiliaTsanira M, Gourounti K. Is the residential combined (psychotherapy plus medication) treatment of patients with severe personality disorder effective in terms of suicidality and impulsivity? J Nerv Ment Dis. 2014 Feb;202(2):138-43. doi: 10.1097/NMD.0000000000000083. PMID 24469526
- [Background] E. Layiou-Lignos, L. Anagnostaki, I. Malogiannis & H. Karamanolaki (2021): The psychoanalytic psychotherapy endeavor in the Greek public sector, Psychoanalytic Psychotherapy, DOI: 10.1080/02668734.2021.1898045
- [Background] Bateman A, Fonagy P. Randomized controlled trial of outpatient mentalization-based treatment versus structured clinical management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1355-64. doi: 10.1176/appi.ajp.2009.09040539. Epub 2009 Oct 15. PMID 19833787
- [Background] Leibniz Institute for Psychology (ZPID). (2019). Open Test Archive: BPDSI-IV. Borderline Personality Disorder Severity Index (Version IV) - deutsche Fassung. Available at: https://www.testarchiv.eu/en/test/9007150κ
- [Background] Bateman, A., Fonagy, P. (2004) Suicide and self-harm inventory. In: Psychotherapy for Borderline Personality Disorder: Mentalization-based treatment. New York, NY: Oxford University Press.
- [Background] Derogatis, L. R. (1993). BSI brief symptom inventory: Administration, scoring, and procedures manual (4th ed.). Minneapolis, MN: National Computer Systems.
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Horowitz, L. M., Alden, L., Wiggins, J., & Pincus, A. (2000). Inventory of Interpersonal Problems Manual. San Antonio, TX: The Psychological Corporation.
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Andrews G, Singh M, Bond M. The Defense Style Questionnaire. J Nerv Ment Dis. 1993 Apr;181(4):246-56. doi: 10.1097/00005053-199304000-00006. PMID 8473876
- [Background] Lenzenweger MF, Clarkin JF, Kernberg OF, Foelsch PA. The Inventory of Personality Organization: psychometric properties, factorial composition, and criterion relations with affect, aggressive dyscontrol, psychosis proneness, and self-domains in a nonclinical sample. Psychol Assess. 2001 Dec;13(4):577-91. PMID 11793901
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Wetzelaer P, Farrell J, Evers SM, Jacob GA, Lee CW, Brand O, van Breukelen G, Fassbinder E, Fretwell H, Harper RP, Lavender A, Lockwood G, Malogiannis IA, Schweiger U, Startup H, Stevenson T, Zarbock G, Arntz A. Design of an international multicentre RCT on group schema therapy for borderline personality disorder. BMC Psychiatry. 2014 Nov 18;14:319. doi: 10.1186/s12888-014-0319-3. PMID 25407009
- [Background] Bremner JD, Bolus R, Mayer EA. Psychometric properties of the Early Trauma Inventory-Self Report. J Nerv Ment Dis. 2007 Mar;195(3):211-8. doi: 10.1097/01.nmd.0000243824.84651.6c. PMID 17468680
- [Background] First MB, Williams JBW, Benjamin LS, Spitzer RL: User's Guide for the SCID-5-PD (Structured Clinical Interview for DSM-5 Personality Disorder). Arlington, VA, American Psychiatric Association, 2015
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). https://doi.org/10.1176/appi.books.9780890425596
- [Derived] Malogiannis I, Anagnostaki L, Aspradaki M, Aristotelidis P, Karambela K, Amperiadou M, Efthymiou V, Kriezi P, Theodoridou I, Stefanatou P, Konstantakopoulos G, Souliotis K, Peppou LE, Giannoulis E. Borderline personality disorder Athens study: a quasi-experimental pragmatic trial for the assessment of a public, psychodynamic, stepped care service for borderline personality disorder patients. Front Psychiatry. 2025 Jul 1;16:1493265. doi: 10.3389/fpsyt.2025.1493265. eCollection 2025. PMID 40666438